CLINICAL TRIAL: NCT00991471
Title: A Cluster Randomized Trial of the Effect of an Physician-Nurse Supplementary Triage Assistance Team (MDRN STAT) on Emergency Department Patient Wait Times
Brief Title: The Effect of an Physician-Nurse Supplementary Triage Assistance Team on Emergency Department Patient Wait Times
Acronym: MDRNSTAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Ivy Cheng, Dr. Ivy Cheng, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 226-2009
Record Dates: First submitted 2009-10-05; First posted 2009-10-08 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Emergencies
Keywords: Emergency Department Wait Times; Physician Nurse at Triage; Overcrowding; CostEffectiveness
MeSH Terms: conditions — Emergencies; Crowding | interventions — Drug Interactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interaction with MDRN STAT (Experimental): Interaction with MDRNSTAT at triage to obtain orders for investigations and/or treatment
  Interventions: Behavioral: Interaction with MDRN STAT
- Control: No MDRNSTAT (Experimental): Control group
  Interventions: Behavioral: No MDRNSTAT

INTERVENTIONS:
Behavioral: Interaction with MDRN STAT — Interaction with MDRNSTAT at triage to obtain orders for investigations and/or treatment
  Arms: Interaction with MDRN STAT
Behavioral: No MDRNSTAT — Standard management of nurse-only triage for assignment of CTAS
  Other Names: Standard triage
  Arms: Control: No MDRNSTAT

SUMMARY:
The primary objective of this study is to investigate whether the introduction of a physician-nurse supplementary triage assessment team (MDRN STAT) is effective in improving time-based performance indicators for wait times. Secondary objectives will examine the quality of patient care and health care worker satisfaction and the cost-effectiveness of the program

DETAILED DESCRIPTION:
In 2007, the Ontario Ministry of Health and Long-term Care (MOHLTC) declared emergency department wait-times a government priority. The crisis of overcrowding and access block has become an international epidemic, affecting developing countries in Europe, North America, and Australasia. The MOHLTC has targeted 23 Ontario hospitals' prolonged wait times. Sunnybrook Health Sciences Center has been selected. Therefore, this is a quality improvement study of patient wait-times and care.

During a 20-week period, the MDRN STAT will be present on randomly chosen weekdays (8:00-16:00) for 50 shifts. Wait-times, such as time from triage time to: physician assessment, stretcher occupation, treatment orders (drugs), investigation orders (laboratory, diagnostic imaging), investigation acquisition (diagnostic imaging), consultation, bed request, discharge from ED (i.e. length of stay (LOS)) time, will be analyzed. In addition, the left-without-being-seen rate (LWBS) and rate of return will be analyzed. These results will be compared to the Ontario wait-time strategy P4R targets, as well as the Canadian Triage Acuity Scale (CTAS guidelines). Economic analysis of this intervention will be done. The hospital will independently perform patient satisfaction surveys. Health care worker satisfaction survey data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients arriving from 8:00-14:30 during a day here a MDRN STAT is assigned

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6300 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the MDRN STAT on emergency department wait times | Time from triage to time of discharge from ED

SECONDARY OUTCOMES:
Cost-Effectiveness of a MDRN STAT in the Emergency Department | 6 months, of 50 MDRN STAT shifts, randomized with non-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ivy Cheng, FRCP, Principal Investigator — Sunnybrook Hospital Emergency Department
Locations (1):
- Sunnybrook Health Sciences Center, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Cheng I, Lee J, Mittmann N, Tyberg J, Ramagnano S, Kiss A, Schull M, Kerr F, Zwarenstein M. Implementing wait-time reductions under Ontario government benchmarks (Pay-for-Results): a Cluster Randomized Trial of the Effect of a Physician-Nurse Supplementary Triage Assistance team (MDRNSTAT) on emergency department patient wait times. BMC Emerg Med. 2013 Nov 11;13:17. doi: 10.1186/1471-227X-13-17. PMID 24207160